CLINICAL TRIAL: NCT07209514
Title: Feasibility and Therapeutic Efficacy Study of Medtronic's DTM-Closed-Loop Integrated SCS Technology for Managing Diabetic Peripheral Neuropathic Pain (DPN)
Brief Title: Medtronic Inceptiv™ Closed-Loop DTM Spinal Cord Stimulation for Painful Diabetic Peripheral Neuropathy
Acronym: MED DPN
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: TriCity Research Center (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIS-25-MTR-001; ERP #14060 (Other Grant/Funding Number: Medtronic)
Record Dates: First submitted 2025-10-01; First posted 2025-10-07 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Diabetic Peripheral Neuropathic Pain (DPN)
Keywords: Diabetic Peripheral Neuropathic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Inceptiv CL DTM SCS (Experimental): Participants undergo a short trial of SCS. Those with a successful trial will receive permanent implantation of the Medtronic Inceptiv SCS with paddle leads. After implant, closed-loop ECAP-guided Differential Target Multiplexed stimulation will be activated and optimized at follow-up visits.
  Interventions: Device: Implantable SCS with Closed Loop mechanism

INTERVENTIONS:
Device: Implantable SCS with Closed Loop mechanism — Participants will be treated with an implantable spinal cord stimulation system programmed to deliver differentially multiplexed targeting pulse program with closed-loop adjustment using evoked compound action potential feedback. All subjects will first undergo a short percutaneous trial phase of spinal cord stimulation. Those who meet trial success criteria will then receive permanent implantation with a paddle lead and the implantable pulse generator. After implantation, closed-loop DTM therapy will be enabled and optimized at each follow-up visit. The goal of the intervention is to evaluate feasibility, safety, and effectiveness of closed-loop DTM spinal cord stimulation in patients with painful diabetic peripheral neuropathy.

SUMMARY:
This study is conducted to evaluate a new way of using spinal cord stimulation (SCS) in people with painful diabetic peripheral neuropathy (DPN). The device used is the Medtronic Inceptiv SCS, which is already approved by the U.S. FDA for treatment of chronic pain. In this study, the system will be programmed to deliver Differential Target Multiplexed (DTM) stimulation with closed-loop feedback using signals from the spinal cord (ECAPs). Up to 25 participants will take part in the study, beginning with a short trial phase and continuing to a permanent implant if the trial is successful. Participants will be followed for 12 months after implant. The main goal is to see whether this therapy can safely and effectively reduce pain in people with diabetic neuropathy. Other measures include physical function, symptom profiles, treatment satisfaction, and monitoring for any side effects.

ELIGIBILITY:
* Inclusion Criteria:

  1. Adults ≥19 years.
  2. Confirmed DPN with EMG evidence of peripheral nerve dysfunction.
  3. Persistent lower-limb neuropathic pain VAS ≥6 for ≥6 months despite prior pharmacologic therapy.
  4. HbA1c ≤8.5% within 3 months prior to enrollment.
  5. No prior SCS/neuromodulation therapy; medically eligible for paddle lead implantation with Inceptiv IPG.
  6. Insurance approval or financial ability to cover SCS therapy; able to consent and comply.
* Exclusion Criteria:

  (a) Non-diabetic neuropathies other conditions contributing to lower-limb pain. (b) Contraindications to surgical implantation.

  (c) History of neurostimulation therapy; active substance abuse or uncontrolled psychiatric illness.

  (d) Pregnancy or plans for pregnancy; known allergy to device materials; inability to provide informed consent.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2027-09-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity on the Visual Analog Scale (VAS, 0-10) from Baseline to 12 Months | Baseline; End of Trial (~7 days after trial lead placement); 1, 3, 6, and 12 months after permanent implant. Primary time point: 12 months.
  Pain intensity is assessed with a 0-10 VAS. Scores are collected at each study visit. The primary endpoint is the change score calculated as 12-month VAS minus baseline VAS; negative values indicate improvement (decrease in pain). Analysis will summarize mean change (SD) and 95% CIs. Additional summaries may include the proportion of participants achieving ≥30% and ≥50% reduction as supportive endpoints.

CONTACTS AND LOCATIONS:
Locations (1):
- Grand Island Pain Relief Center, Grand Island, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Undecided